CLINICAL TRIAL: NCT03492541
Title: Evaluation of the Clinical Efficacy and Tolerability of SYSTANE Complete in Adult Patients With Dry Eye Disease Following Topical Ocular Use for 4 Weeks: A Multicenter Trial
Brief Title: Study of Efficacy and Tolerability of SYSTANE Complete in Patients With Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDMGD0012401
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Dry Eye Disease
Keywords: mixed dry eye; aqueous-deficient dry eye; lipid-deficient dry eye; evaporative dry eye; tear film; eye drops; artificial tears; lipid layer; eye symptoms; meibomian gland dysfunction; MGD; SYSTANE; SYSTANE Complete; nanoemulsion
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYSTANE Complete (Experimental): Propylene glycol-based eye drops, 1 drop in each eye twice a day (BID) (morning and evening) for 28 days. Patients can administer additional doses in between the scheduled daily doses as needed
  Interventions: Other: Propylene glycol-based eye drops

INTERVENTIONS:
Other: Propylene glycol-based eye drops — Nano-emulsion ocular lubricant
  Other Names: SYSTANE® Complete

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness and tolerability of SYSTANE® Complete in adult patients with dry eye disease. Fluorescein-stained tear film break-up time (TFBUT) will be evaluated as the primary objective.

DETAILED DESCRIPTION:
Patients will attend 4 scheduled visits: Screening Visit (Day -7 to Day 0), Visit 1/Baseline Visit (Day 1), Visit 2 (Day 14) and Visit 3 (Day 28).

ELIGIBILITY:
Inclusion Criteria:

* Must have TFBUT of ≤ 5 seconds in at least one eye at Screening visit.
* Must have best corrected visual acuity (BCVA) of ≥ 20/80 (or ≥ 55 letters score or ≥ 0.6 early treatment diabetic retinopathy study (ETDRS) log of the minimum angle of resolution (LogMAR) value) in both eyes at the Screening visit.
* Must be willing to discontinue use of all artificial tear supplements and use only the study product as directed for the entire study duration.

Exclusion Criteria:

* History of hypersensitivity to the study drug or any of its excipients or to drugs of similar chemical classes.
* Use of any topical ocular medication preserved with benzalkonium chloride or other products known to be toxic to the tear film lipid layer within 1 month prior to the Screening visit.

Other protocol-specified inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Tear Film Break-up Time (TFBUT) at Day 14 | Baseline, Day 14
  TFBUT will be assessed using fluorescein, an ocular staining dye

SECONDARY OUTCOMES:
Change from baseline in dry eye symptom score at Day 1 | Baseline, Day 1
  As reported by the patient using a Likert scale post drop instillation
Soothing sensation score | Day 1
  As reported by the patient using a Likert scale post drop instillation
Tolerability assessment score | Day 1
  As reported by the patient using an assessment questionnaire post drop instillation
Change from baseline in ocular discomfort at Day 14 | Baseline, Day 14
  As reported by the patient using a Visual Analogue Scale (VAS)
Change from baseline in corneal staining score at Day 28 | Baseline, Day 28
  Assessment of ocular staining using staining dye under a slit lamp
Change from baseline in response to the revised IDEEL questionnaire at Day 28 | Baseline, Day 28
  As reported by the patient using a subjective questionnaire
Change from baseline in EQ-5D-5L score(s) at Day 28 | Baseline, Day 28
  As reported by the patient using a validated questionnaire
Change from baseline in TFBUT at Day 28 | Baseline, Day 28
  TFBUT will be assessed using fluorescein, an ocular staining dye

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Pharmaceuticals, Study Director — Alcon Research
Locations (4):
- United States (2):
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, Norfolk, Virginia
- Investigative Site, Valladolid, Castille and León, Spain
- Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No